CLINICAL TRIAL: NCT03319329
Title: Metabolic Determinants Of Resting Energy Expenditure Among Mechanically Ventilated Critically Ill Patients In Malaysian Tertiary Hospital
Brief Title: Metabolic Determinants Of Resting Energy Expenditure Among Mechanically Ventilated Critically Ill Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Tah Pei Chien, Department of Anesthesiology, Faculty of Medicine, University of Malaya
Other Study IDs: 20161024-4407
Record Dates: First submitted 2017-09-23; First posted 2017-10-24 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness | interventions — Calorimetry, Indirect

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- critically ill adult patients: Part I: A cross-sectional study to compare validity of several predictive equations used to predict REE in critically ill adult patients for staying ≤ 5 days, 6 - 10 days and > 10 days by using indirect calorimetry (IC) as the reference standard.
  Part II: To develop predictive equation for the estimation of energy requirement by identifying variables that might influence REE of mechanically ventilated critically ill patients.
  Part III: To validate the newly developed predictive equation for the estimation of energy requirement by using Ten fold cross-validation approach
  Interventions: Device: Indirect Calorimetry

INTERVENTIONS:
Device: Indirect Calorimetry — REE measurements were using IC (Cosmed, Quark RMR 2.0, Indirect Calorimetry Lab, Italy). A standard protocol for conducting the measurement was followed (Schlein & Coulter, 2014);(P. Singer & Singer, 2016); (Taku Oshima et al., 2016). Before each measurement, the metabolic monitor was allowed to warm up for 30 min, and then gas and flowmeter calibrations were performed by an experienced dietitian or healthcare professional. The REE was recorded after a 30 min non-fasting steady state according to RMR protocol and manufacturer instructions.

SUMMARY:
Currently there are no study related to Indirect Calorimetry (IC) has been done among hospitalised Malaysian ICU adult patients with its racial mix. The aim of this study is to perform a cross-sectional study in Malaysian critically ill patients to determine metabolic determinants that might influence resting energy expenditure (REE) and to develop predictive equation for the estimation of energy requirement using the regression based approach to increase the accuracy in calorie prescriptions. In addition, expected outcome of this study is to determine which equations have clinical usefulness among Malaysian adult critically ill patients and hope to introduce into routine clinical practice in the future if IC is not available.

DETAILED DESCRIPTION:
Nutrition provision in the clinical setting relies heavily on the accurate estimation of energy and protein requirements. This can be done in a quick and inexpensive manner via the use of predictive equations. Some of the most popularly used predictive equations such as the Harris-Benedict equation and the Mifflin-St. Jeor equation have been widely applied within the clinical setting to estimate energy requirements among mechanically ventilated critically ill patients. However, these existing equations were not specially developed for a population with disease, as the equations were derived from a pool of healthy Caucasian adults. In addition, most of the equations for critically ill patients such as the Penn State equation, Faisy equation and Raurich Equation developed and validated among Caucasian in western country and not among Asian population. Therefore, their accuracy in predicting energy requirement is questionable when applied within Malaysian mechanically ventilated critically ill patients with its racial mix.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged over 18 years old
2. Critically ill patients with mechanically ventilated
3. Expected to have an ICU stay of more than 5 days
4. Patients had implemented for continuous enteral or parenteral nutrition support.

Exclusion Criteria:

1. Requirement for inspired oxygen content (FiO2) greater than 0.6
2. Patients on high frequency ventilation
3. Patients with chest tubes that leak air
4. Patients with incompetent tracheal cuff
5. Patients inhaled nitric oxide therapy
6. Patients receiving intermittent hemodialysis and continuous renal replacement therapy (CRRT) during IC measurement
7. Patients with pregnancy
8. Patients with burn injury
9. Patients infected with human immunodeficiency virus (HIV)
10. Patients with severe liver disease (Child-Pugh score C)
11. Patients with post open heart surgery
12. Patients with paraplegia and quadriplegia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients with mechanically ventilated
Sampling Method: Probability Sample
Enrollment: 314 (Estimated)
Dates: Start 2017-02-13 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants measured resting energy expenditure for the development of predictive equations | 24 months
  predictive equations for the estimation of energy requirement among mechanically ventilated critically ill patients among Malaysian population.

SECONDARY OUTCOMES:
The validity of several predictive equations by using Intraclass Correlation Coefficient (ICC) test | 24 months
  predictive equations used to predict REE in critically ill adult patients among Malaysian population by using indirect calorimetry (IC) as the reference standard.
Determine metabolic determinants | 24 months
  metabolic determinants that might influence resting energy expenditure among mechanically ventilated critically ill patients.
The best regression equation model | 24 months
  Regression equation model for predicting energy requirement of mechanically ventilated critically ill patients.
Determine and compare REE measured by IC among mechanically ventilated critically ill patients | 24 months
  during early phase (staying ≤ 5 days), late phase (staying 6-10 days) and chronic phase (staying > 10 days) in ICU.
The association of REE in critically ill patients with clinical outcome | 24 months
  Clinical outcome are hospital mortality and ICU mortality in 28 days and 60 days, length of mechanical ventilation in hours, duration of ICU stay in days and infectious complications such as Hospital acquired infection.
The association of REE in critically ill patients with quality of life | 24 months
  Questionnaire SF-36v2 Health Survey to measure quality of life for critically ill patients.
The association of REE in critically ill patients with nutrition risk | 24 months
  NUTRIC score to quantify the nutrition risk of critically ill patients developing adverse events
The energy and protein adequacy in relation to patient outcome. | 24 months
  Energy and protein adequacy in terms of Energy/Nitrogen ratio in relation to patient outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Pei Chien Tah, Principal Investigator — UNIVERSITY OF MALAYA MEDICAL CENTRE
Locations (1):
- University of Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia

REFERENCES:
- [Derived] Tah PC, Poh BK, Kee CC, Lee ZY, Hakumat-Rai VR, Mat Nor MB, Kamarul Zaman M, Majid HA, Hasan MS. Do we need different predictive equations for the acute and late phases of critical illness? A prospective observational study with repeated indirect calorimetry measurements. Eur J Clin Nutr. 2022 Apr;76(4):527-534. doi: 10.1038/s41430-021-00999-y. Epub 2021 Aug 30. PMID 34462560